CLINICAL TRIAL: NCT02218060
Title: Coronary CT Angiography Using a Novel 3rd Generation Dual-Source CT System: Diagnostic Performance and Potential for Reduction in Radiation Dose and Contrast Material Requirement
Brief Title: Coronary CT Angiography Using a Novel 3rd Generation Dual-Source CT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, U. Joseph Schoepf, MD, Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Force Cardiac
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Force (Experimental): Patients receiving coronary CT angiography on the SOMATOM Force before clinically indicated cardiac catheterization or after clinically indicated nuclear stress test
  Interventions: Procedure: Coronary CT angiography on SOMATOM Force
- Control (Other): Patients who have already received comparable CT examinations on current routine 2nd generation dual-source CT systems
  Interventions: Procedure: Previous coronary CT angiography on 2nd generation CT scanner

INTERVENTIONS:
Procedure: Coronary CT angiography on SOMATOM Force — Coronary CT angiography using iodinated contrast; metoprolol and/or nitroglycerin may also be administered on a per-patient basis
  Arms: Force
Procedure: Previous coronary CT angiography on 2nd generation CT scanner — Clinically indicated coronary CT angiography previously performed on a 2nd generation CT scanner
  Arms: Control

SUMMARY:
Coronary CT angiography is used to examine the coronary arteries in a non-invasive way when a patient is suspected of having coronary artery disease. The test, however, requires relatively high levels of radiation, which have been linked to DNA damage and cancer, and the use of contrast material, which can affect kidney function. The SOMATOM Force, a new third-generation CT scanner manufactured by Siemens, was recently installed at MUSC and holds the potential to obtain quality images while also reducing radiation dose and contrast material. This study aims to test the diagnostic ability of the SOMATOM Force in detecting coronary artery disease and also see if radiation dose and contrast material are reduced compared to the previous 2nd generation scanners. It is suspected that the Force will provide clinical quality images while decreasing radiation dose and contrast material required.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18-90 years of age.
* Subject must have been referred for a clinically indicated cardiac catheterization or nuclear cardiac perfusion study.
* Subject must provide written informed consent prior to any study-related procedures being performed.
* Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

* Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

  * By testing (urine βHCG) within 24 hours before contrast agent administration, or
  * By surgical sterilization, or
  * Post menopausal, with minimum one (1) year history without menses.
* Subject has an acute psychiatric disorder or is cognitively impaired.
* Subject is using or is dependent on substances of abuse.
* Subject is unwilling to comply with the requirements of the protocol.
* Subject has decreased renal function (eGFR <45)
* Subject has an allergy against iodinated contrast agents.
* Subject is in acute unstable condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Radiation dose and contrast material | one year
  To determine the potential for reductions in radiation dose and contrast material requirements by performing coronary CT angiography at low tube potential with the new CT system.

SECONDARY OUTCOMES:
Diagnostic accuracy | one year
  To determine the diagnostic accuracy of coronary CT angiography performed with the new CT system using coronary catheterization or nuclear myocardial perfusion imaging as reference standards.

CONTACTS AND LOCATIONS:
Overall Officials: U. Joseph Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Ashley River Tower, Charleston, South Carolina, United States